CLINICAL TRIAL: NCT00463957
Title: The Pharmacological Basis for the Increase in Visual Time Constants Induced by Single Oral Doses of Sildenafil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cambridge (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: REC 06/Q0108/200
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2007-04

CONDITIONS: Erectile Dysfunction
Keywords: sildenafil; tadalafil; phosphodiesterase; visual persistence; reaction time
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sildenafil
Drug: tadalafil
Drug: placebo

SUMMARY:
Sildenafil and similar drugs have been used for several years to treat erectile dysfunction. It has been noticed that in some people, sildenafil causes a subtle increase in the length of time that visual images that we see are retained by the retina. It is thought that this might be due to an effect of sildenafil on inhibiting an enzyme called phosphodiesterase type 6 (PDE6) which is present in the retina. By giving single oral doses of sildenafil and a similar drug called tadalafil which has less effect on PDE6, we hypothesise that this is the mechanism of the change in vision caused by sildenafil. By performing computerised visual test, we plan to compare the effects of sildenafil, tadalafil and placebo tablets on vision in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18-55 years

Exclusion Criteria:

* Significant medical or psychiatric illness
* Cardiac disease
* Hyper or hypotension
* Renal disease
* Liver disease
* Stroke
* Sickle cell anaemia
* Multiple myeloma
* Leukaemia
* Bleeding disorders
* Peyronie's disease
* Priapism
* Subjects receiving prescribed medications
* Subjects with known visual abnormalities other than refractive errors, including retinitis pigmentosa, optic neuropathy

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2006-08

PRIMARY OUTCOMES:
visual persistence
reaction time

CONTACTS AND LOCATIONS:
Overall Officials: Morris J Brown, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom